CLINICAL TRIAL: NCT05602519
Title: The Analgesic Efficacy and Safety of Oxycodone Hydrochloride Versus Fentanyl After Total Hip Arthroplasty: A Randomized Triple-Blind Trial
Brief Title: The Analgesic Efficacy of Oxycodone Hydrochloride Versus Fentanyl After Total Hip Arthroplasty:
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 00012367-22-010-005
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Total Hip Arthroplasty; The Analgesic Efficacy
Keywords: Oxycodone Hydrochloride; Fentanyl
MeSH Terms: interventions — Propofol; Rocuronium; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group fentanyl (Active Comparator): Patients will receive 50 ug of fentanyl 20 min before the end of surgery.
  Interventions: Drug: propofol, rocuronium and fentanyl
- Group oxycodone (Active Comparator): Patients will receive 4 mg of oxycodone 20 min before the end of surgery.
  Interventions: Drug: propofol, rocuronium and fentanyl

INTERVENTIONS:
Drug: propofol, rocuronium and fentanyl — In fentanyl group (36 patients), 50 ug of fentanyl, and in oxycodone group, 4 mg of oxycodone will be administered 20 minutes before the end of the surgery, in triple blind manner.

SUMMARY:
Oxycodone showed similar or superior analgesic effects than fentanyl and was proposed as an alternative for fentanyl for pain control in the postoperative period. However, it was mainly directed to control visceral pain, due to the mediation of analgesic effects by the kappa receptors. However, few studies compared the oxycodone to fentanyl for postoperative pain relief in patients undergoing total hip arthroplasty (replacement). Therefore, we established this randomized study to compare the efficacy of oxycodone and fentanyl for relief of postoperative pain after total hip arthroplasty (replacement).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 28-62 years old,
* Both genders, American Society of Anesthesiologists (ASA) physical status classification I or II who scheduled for elective total hip surgery.

Exclusion Criteria:

* Patients with history of any kind of drug allergy.
* drug abuse.
* psychological or other emotional problems,
* renal and hepatic chronic disease.

Ages: 28 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Improving A post-anesthesia care unit (PACU) pain score. | 48 hours
  The visual analogue scale (VAS) will be used for assessment of postoperative pain severity (0 for no pain and 10 for the most severe pain).

SECONDARY OUTCOMES:
Hemodynamics | 48 hours
  Mean arterial blood pressure and heart rate will be recorded at baseline and every 5 min till the end of procedure.
Postoperative side effects | 48 hours
  Any side effects will be documented. Postoperative nausea and vomiting (if occurred) will be treated by intravenous administration of metoclopramide (10mg).
Postoperative consumption of opioid | 48 hours postoperatively
  The overall dose of fentanyl administrated in the first 48 postoperative hours will be documented at 6, 12, 24 and 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Facualty of Medicine (Damietta), Al Azhar University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with a reasonable request with corresponding author.
Supporting Information: Study Protocol, SAP